CLINICAL TRIAL: NCT04354467
Title: Assessment of Urinary Neutrophil Gelatinase-Associated Lipocalin (NGAL) Ito Predict Acute Kidney Injury (AKI) in the NICU in Infants Receiving Multiple Nephrotoxic Medications (NICU NINJA NGAL)
Brief Title: Assessment of Urinary Neutrophil Gelatinase-Associated Lipocalin to Predict AKI in the NICU
Status: Completed | Type: Observational
Sponsor: University of Alabama at Birmingham (Other)
Collaborators: Children's Hospital Medical Center, Cincinnati (Other)
Responsible Party: Principal Investigator, David Askenazi, Principal Investigator, University of Alabama at Birmingham
Other Study IDs: 300000362
Record Dates: First submitted 2020-04-16; First posted 2020-04-21 (Actual); Last update posted 2024-01-05 (Actual); Status verified 2024-01

CONDITIONS: Acute Kidney Injury; Nephrotoxicity; Neonatal
MeSH Terms: conditions — Acute Kidney Injury

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Urine
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Neonates exposed to Nephrotoxic Medications: Neonates exposed to Nephrotoxic Medications as defined by the NINJA inclusion criteria
  Interventions: Diagnostic Test: urine neutrophil gelatinase -associated lipocalin

INTERVENTIONS:
Diagnostic Test: urine neutrophil gelatinase -associated lipocalin — urine biomarker is measured and batched procesessed
  Other Names: urine NGAL

SUMMARY:
Nephrotoxic medication (NTMx) exposure is one of the most commonly cited causes of acute kidney injury (AKI) in hospitalized children, and is the primary cause of AKI in 16% of cases. Through initial work at UAB/Children's of Alabama Hospital, NTMx exposure was found to be potentially modifiable and the associated AKI is an avoidable adverse safety event. Currently, only serum Creatinine monitoring is available to monitor for NTMx-associated AKI. The hypothesis of this NINJA NGAL study is that urine NGAL is highly sensitive to detect NTMx-associated AKI. UAB/Children's of Alabama is bringing urine NGAL measurement to the infants in the NICU to detect NTMX-associated AKI.

DETAILED DESCRIPTION:
Nephrotoxic medication-induced acute kidney injury (NTM-AKI) is a relevant yet underdiagnosed morbidity in the neonatal intensive care unit (NICU).

Up to 87% of very low birth weight infants are exposed to at least one nephrotoxic medication (NTM). NTM-AKI is associated with poor short and long-term outcomes.

Presently, no treatments exist for AKI beyond supportive care.

ELIGIBILITY:
Inclusion Criteria:

* all NICU inpatients under 1 year of age; greater than 4 days of age that are

  * Receiving 3 or more nephrotoxic medications on the same day OR
  * Receiving 3 or more days of an intravenous aminoglycoside or vancomycin

Exclusion Criteria:

* Less than 4 days of age

  * Currently being treated for a urinary tract infection
  * Presence of an acute kidney injury prior to enrollment

Max Age: 1 Year | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Admitted to Neonatal Intensive Care Unit
Sampling Method: Non-Probability Sample
Enrollment: 148 (Actual)
Dates: Start 2019-01-28 (Actual); Primary Completion 2020-12-30 (Actual); Study Completion 2023-12-30 (Actual)

PRIMARY OUTCOMES:
Percentage of patients with elevated urine NGAL | Daily for one week after meeting criteria for nephrotoxic medication exposure
  NGAL is an early, sensitive, non-invasive urine biomarker for AKI.

CONTACTS AND LOCATIONS:
Overall Officials: David Askenazi, Principal Investigator — University of Alabama at Birmingham
Locations (2):
- United States (2):
  - Children's of Alabama, Birmingham, Alabama
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio

IPD SHARING:
Plan to Share IPD: Yes
upon request
Supporting Information: Study Protocol, CSR
Time Frame: in 2025 for 4 years

REFERENCES:
- [Result] Stoops C, Gavigan H, Krallman K, Anderson N, Griffin R, Slagle C, House S, Goldstein SL, Askenazi DJ. The Utility of Urinary NGAL as an Alternative for Serum Creatinine to Detect Acute Kidney Injury in Infants Exposed to Nephrotoxic Medications in the Neonatal Intensive Care Unit. Neonatology. 2024;121(2):203-212. doi: 10.1159/000535322. Epub 2023 Dec 27. PMID 38151013